CLINICAL TRIAL: NCT03616938
Title: Impact of Newly Infant Chest Compression Technique on Hemodynamic Effect During CPR: A Multicenter Randomized Crossover Experimental Study
Brief Title: Infant Chest Compression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Łukasz Szarpak (Other)
Collaborators: Wroclaw Medical University (Other)
Responsible Party: Sponsor-Investigator, Łukasz Szarpak, Associate Professor, Lazarski University
Organization: Lazarski University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NLS_2018_UL
Record Dates: First submitted 2018-07-31; First posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Cardiac Arrest; Infant; Simulation
Keywords: cardiopulmonary resuscitation; chest compression; medical simulation; randomization; quality
MeSH Terms: conditions — Heart Arrest | interventions — Cardiopulmonary Resuscitation

STUDY DESIGN:
Who Masked: Participant
Masking Description: study participant had no insight on the simulator or a cardio-monitor display
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- the two finger chest compression technique (Experimental): Two finger technique (TFT): the pediatric thorax is compressed with the tips of two fingers and is recommended for lone rescuer during infant cardiopulmonary resuscitation by international resuscitation guidelines
  Interventions: Procedure: Cardiopulmonary resuscitation
- the two thumb chest compression technique (Experimental): Two thumb technique (TTHT): the two thumbs of the rescuer are placed over the lower third of the sternum, with the fingers encircling the torso and supporting the back. This technique is recommended for two rescuers during infant CPR by international CPR guidelines
  Interventions: Procedure: Cardiopulmonary resuscitation
- the new two thumb chest compression technique (Experimental): 'new two-thumb technique' (nTTT): this technique consists in using two thumbs directed at the angle of 90° to the chest while closing the fingers of both hands in a fist
  Interventions: Procedure: Cardiopulmonary resuscitation

INTERVENTIONS:
Procedure: Cardiopulmonary resuscitation — 2-min cycle of cardiopulmonary resuscitation accorind to the American Heart Association 2015 guidelines

SUMMARY:
our aim was to quantitatively compare the quality of chest-compression of the new two thumb chest compression (nTTT) versus the current standard techniques: two finger technique (TFT), two thumb technique (TTHT) as defined by systolic-, diastolic-, mean arterial- and pulse-pressures. Our hypothesis is that nTTT generates higher arterial blood pressures compared to the established TFT and TTHT in an infant manikin model.

DETAILED DESCRIPTION:
To simulate the scenario of infant CPR, an ALS Baby trainer manikin (Laerdal Medical, Stavanger, Norway) simulating a 3-month-old infant. The manikin was connected with a fixed-volume arterial system attached to a monitor (Draeger Infinity® Delta; Draegerwerk AG & Co. KGaA, Luebeck, Germany) via an arterial pressure transducer (Edward Lifesciences: TruWave Disposable Pressure Transducer; Irvine, CA, USA). The arterial circuit composed of a 50-mL bag of normal saline solution (air removed) attached to the manikin chest plate and connected to the transducer with a 20-gauge intravenous catheter and tubing. The manikin was placed on a high adjustable hospital stretcher. The bed was leveled to the iliac crest of each rescuer for standardization. The manikin was previously intubated and ventilation was performed using a resuscitator bag.

ELIGIBILITY:
Inclusion Criteria:

* nurses
* give voluntary consent to participate in the study

Exclusion Criteria:

* not meet the above criteria
* wrist or low back diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2018-07-28 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
systolic blood pressure (SBP) | 1 day
  The manikin was connected with a fixed-volume arterial system attached to a monitor (Draeger Infinity® Delta; Draegerwerk AG & Co. KGaA, Luebeck, Germany) via an arterial pressure transducer (Edward Lifesciences: TruWave Disposable Pressure Transducer; Irvine, CA, USA). The arterial circuit composed of a 50-mL bag of normal saline solution (air removed) attached to the manikin chest plate and connected to the transducer with a 20-gauge intravenous catheter and tubing.

SECONDARY OUTCOMES:
diastolic blood pressure (DBP) | 1 day
  The manikin was connected with a fixed-volume arterial system attached to a monitor (Draeger Infinity® Delta; Draegerwerk AG & Co. KGaA, Luebeck, Germany) via an arterial pressure transducer (Edward Lifesciences: TruWave Disposable Pressure Transducer; Irvine, CA, USA). The arterial circuit composed of a 50-mL bag of normal saline solution (air removed) attached to the manikin chest plate and connected to the transducer with a 20-gauge intravenous catheter and tubing.
mean arterial pressure (MAP) | 1 day
  The manikin was connected with a fixed-volume arterial system attached to a monitor (Draeger Infinity® Delta; Draegerwerk AG & Co. KGaA, Luebeck, Germany) via an arterial pressure transducer (Edward Lifesciences: TruWave Disposable Pressure Transducer; Irvine, CA, USA). The arterial circuit composed of a 50-mL bag of normal saline solution (air removed) attached to the manikin chest plate and connected to the transducer with a 20-gauge intravenous catheter and tubing.

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Szarpak, PhD, Study Director — Lazarski University
Locations (1):
- Faculty of Medicine, Lazarski University, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided
Data will be available from the principal investigator

REFERENCES:
- [Background] Smereka J, Szarpak L, Ladny JR, Rodriguez-Nunez A, Ruetzler K. A Novel Method of Newborn Chest Compression: A Randomized Crossover Simulation Study. Front Pediatr. 2018 May 29;6:159. doi: 10.3389/fped.2018.00159. eCollection 2018. PMID 29896467
- [Background] Ladny JR, Smereka J, Rodriguez-Nunez A, Leung S, Ruetzler K, Szarpak L. Is there any alternative to standard chest compression techniques in infants? A randomized manikin trial of the new "2-thumb-fist" option. Medicine (Baltimore). 2018 Feb;97(5):e9386. doi: 10.1097/MD.0000000000009386. PMID 29384839
- [Background] Smereka J, Szarpak L, Smereka A, Leung S, Ruetzler K. Evaluation of new two-thumb chest compression technique for infant CPR performed by novice physicians. A randomized, crossover, manikin trial. Am J Emerg Med. 2017 Apr;35(4):604-609. doi: 10.1016/j.ajem.2016.12.045. Epub 2016 Dec 19. PMID 28040386